# Evaluation of quality of vision and visual outcomes with bilateral implantation of the Clareon PanOptix intraocular lens

An investigator-initiated clinical trial

#### 1. TITLE PAGE

Protocol Number: THN-22-001

Amendment Number Version 1.0

IRB / ERC Salus IRB

2111 West Braker Lane, Suite 400

Austin, Texas 78758

Sponsor Name & Address: Thomas Newsom, MD

Newsom Eye & Laser Center

4211 US Hwy 27 N Sebring, FL 33870 (863)-385-1544

(funding only, this is an investigator-initiated study

*IIT # 72606713*)

Alcon

6201 South Freeway,

Fort Worth, TX 76134-2099, USA

Test Articles: The Clareon<sup>TM</sup> PanOptix<sup>TM</sup> Trifocal (toric and non-toric models)

Investigator: Thomas Newsom, MD

Newsom Eye & Laser Center

4211 US Hwy 27 N Sebring, FL 33870 (863-385-1544)

#### 2. INVESTIGATOR AGREEMENT

I confirm that I have read and that I understand this protocol entitled "Evaluation of quality of vision and visual outcomes with bilateral implantation of the Clareon PanOptix intraocular lens", and understand the use of the study products. I agree to conduct this study in accordance with the requirements of this protocol and also protect the rights, safety, privacy, and well-being of study subjects in accordance with the following:

- The ethical principles that have their origin in the Declaration of Helsinki.
- All applicable laws and regulations, including, without limitation, data privacy laws and regulations.
- Regulatory requirements for reporting serious adverse events defined in Section 13 of this protocol.

| Signature of Investigator (Date) |
|-----------------------------------|
| Investigator Name (print or type) |
| Investigator's Title |
| Name of Facility |
| Location of Facility (City) |

#### 3. GENERAL INFORMATION

Objective To evaluate visual outcomes and quality of vision following

bilateral implantation of the Clareon PanOptix intraocular lens

(IOL) targeted for emmetropia.

The hypothesis is that the Clareon<sup>TM</sup> PanOptix<sup>TM</sup> Trifocal IOL will provide good overall quality of vision and visual outcomes.

Test Article(s) The Clareon<sup>TM</sup> PanOptix<sup>TM</sup> Trifocal (toric and non-toric models)

Control Article(s) None.

Sample size 70 eyes of 35 subjects

Study Population Subjects  $\geq$ 40 years of age presenting for cataract surgery who are

interested in reducing their dependence on spectacles at all distances, and who are appropriate candidates for trifocal lens

implantation.

Number of sites One

Study Design Prospective, non-randomized, single-arm study.

Masking None

Variables Primary: Binocular distance-corrected near (40 cm) visual

acuity), 1 and 3-months postop

#### Secondary:

- Bilateral visual acuity outcomes (uncorrected and bestdistance-corrected) at distance (6m), intermediate (60 cm), and near (40 cm), 1 and 3-months postop
- Manifest refraction (residual spherical equivalent refraction, residual sphere, and residual astigmatism), 1 and 3-months postop
- Binocular, distance corrected defocus curve at 3 month post-operatively, using standard parameters: (+1.00 to -3.00 in 0.50D except +0.50 to -0.50 in 0.25D).
- Questionnaire for visual disturbance scores (QUVID)

• Patient satisfaction questionnaire scores (IOLSAT)

# **Exploratory:**

• Binocular DCNVA at 33cm, 1 and 3-months post-operatively.

Duration / Follow-up Preoperative to 3 months postoperative

The study will be registered with clinicaltrials.gov.

The study will be conducted in compliance with the protocol, GCP and applicable regulatory requirements

# 4. TABLE OF CONTENTS 9.1. Informed Consent / Subject enrollment .......9 9.2. Visits and Examinations.......9 12. CONFIDENTIALITY/PUBLICATION OF THE STUDY .......14

| 13.5. Safety Analyses | 18 |
|----------------------------------------------------------------|----|
| 14. GCP, ICH and ETHICAL CONSIDERATIONS | 18 |
| 14.1 Confidentiality | 18 |
| 15. STANDARD EVALUATION PROCEDURES | 19 |
| Table 15.1. Proposed Visits and Study Assessments | 19 |
| 16. DATA CONFIDENTIALITY | 19 |
| 17. FINANCIAL AND INSURANCE INFORMATION/STUDY RELATED INJURIES | 20 |
| 18. STUDY ENDPOINT CRITERIA | 20 |
| 18.1. Patient Completion of Study | 20 |
| 18.2. Patient Discontinuation | 20 |
| 18.3. Patient Termination | 20 |
| 18.4. Study Termination | 20 |
| 18.5. Study Completion | 20 |
| 19. SUMMARY OF RISKS AND BENEFITS | 21 |
| 19.1. Summary of risks | 21 |
| 19.2. Summary of benefits | 21 |
| REFERENCES | 21 |

#### 5. INTRODUCTION

Previous studies have shown that the AcrySof® PanOptix<sup>TM</sup> IOL (Alcon Vision LLC, Fort Worth, Texas, USA) provides good visual outcomes for patients at distance, intermediate and near.<sup>1,2</sup> We are interested in determining the binocular distancecorrected near (40 cm) visual acuity when the Clareon<sup>TM</sup> PanOptix<sup>TM</sup> IOL is implanted bilaterally.

# 6. OBJECTIVE(S)

To evaluate visual outcomes and quality of vision following bilateral implantation of the Clareon PanOptix intraocular lens (IOL) targeted for emmetropia.

#### 7. SUBJECTS

#### 7.1. Subject Population

Eligible test subjects will be presenting for cataract surgery who are interested in a reduced dependence on spectacles for near, intermediate and distance vision, and who are considered appropriate candidates for trifocal lens implantation.

A total of 70 eyes of 35 subjects at one site will be enrolled. Both eyes of a subject must be enrolled. Subjects must meet the inclusion criteria. Prior to enrollment, subjects will be provided information on the study and asked to sign a patient information and consent form to participate. The patient information and consent form will be approved by an appropriate ethics committee.

#### 7.2. Inclusion Criteria

Subjects are eligible for the study if they meet the following criteria:

**Note:** Ocular criteria must be met in both eyes.

- Presenting for uncomplicated bilateral cataract surgery and have an interest in spectacle independence using a trifocal IOL
- Meet the requirements for on-label implantation of the trifocal IOL
- Gender: Males and Females.
- Age: 40 or older.
- Willing and able to provide written informed consent for participation in the study.
- Willing and able to comply with scheduled visits and other study procedures.
- Have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error and cataract).
- Expected visual potential of 20/25 Snellen (0.10 logMAR) or better in each eye.

• All eyes will be in the range of availability for Clareon PanOptix IOL and Clareon PanOptix Toric IOL. For cylinder below the Toric IOL indication (T3), an LRI will be used during surgery.

#### 7.3. Exclusion Criteria

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

- Patients with any corneal pathology (including corneal dystrophies, scaring, severe dry eye syndrome, irregular astigmatism, HOA) limiting or affecting visual potential.
- Patients with previous corneal refractive surgery.
- Patients with pre-existing ocular pathology, including maculopathy, ARMD, ERM, prior RD, and glaucoma limiting or affecting visual potential.
- Subjects who have an unstable acute or chronic disease or illness that would confound the results of this investigation (*e.g.*, immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect postoperative visual acuity.
- Participation in any investigational drug or device trial within the previous 30 days prior to the start date of this trial (or currently participating).

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

#### 8. STUDY DESIGN

#### 8.1. Study Design

This study is a single-arm unmasked clinical evaluation study of binocular distance-corrected near (40 cm) visual acuity after successful bilateral cataract surgery. Subjects will be assessed pre-operatively, operatively and at 1 day, 1 month and 3 months post-operatively. Clinical evaluations will include administration of a visual disturbance questionnaire (QUVID), and a satisfaction questionnaire (IOLSAT), as well as measurement of bilateral visual acuity and manifest refraction.

The primary outcome measure will be the binocular distance-corrected near (40 cm) visual acuity at 1 and 3 months postoperative.

Secondary outcome measures are as follows:

- Bilateral visual acuity outcomes (uncorrected and best-distance-corrected) at distance (6m), intermediate (60 cm), and near (40 cm), 1 and 3-months postop
- Manifest refraction (residual spherical equivalent refraction, residual sphere, and residual astigmatism), 1 and 3-months postop
- Binocular, distance corrected defocus curve at 3 month post-operatively, using standard parameters: (+1.00 to -3.00 in 0.50D except +0.50 to -0.50 in 0.25D).
- Questionnaire for visual disturbance scores (QUVID)
- Patient satisfaction questionnaire scores (IOLSAT)

Exploratory outcome measures are as follows:

• Binocular DCNVA at 33cm, 1 and 3-months post-operatively

#### 8.2. Methods Used to Minimize Bias

As a single-arm study there is no expected bias. Patient selection will be based on the patient's interest and the surgeon's opinion as to whether they are a suitable candidate for trifocal or trifocal toric IOL implantation.

The measurement of visual acuity will be conducted in a systematic fashion to minimize bias. Individuals conducting visual acuity measures will be instructed to perform the same testing in the same fashion for all subjects, with the same level of encouragement to subjects. Questionnaire instructions will be provided to all patients in a similar manner.

All data collection will be completed through provided Case Report Forms (CRFs) or computer files generated by automated test equipment. All site personnel involved in the study will be trained in regard to conducting study-specific procedures.

#### 9. STUDY PROCEDURE

# 9.1. Informed Consent / Subject enrollment

No subject will be enrolled into the study who does not meet the inclusion/exclusion criteria and does not sign the current approved informed consent document. Informed consent will be obtained prior to collecting any data for the study. The original signed documents will be maintained by the investigator as a permanent part of the subject's medical records. A signed copy will be provided to the subject.

#### 9.2. Visits and Examinations

Subjects will participate in seven study visits, one eye per visit for bilateral surgery. Visits will include an uptake visit, two operative visits, and 4 total postoperative visits (Visit numbers 1-5 below). The visit schedule, complete with window and associated

CRF forms, are displayed in Table 9.2-1. Details of each study visit, including testing to be conducted, are provided below.

Table 9.2-1. Visit Schedule

| Visit<br>Number | Visit Name | Visit Window | CRF<br>Number |
|---|---|---|---|
| 1 | Preoperative | -30 to 0 days from surgery | 1 |
| 2,2a | Operative | 0 from surgery | 2,2a |
| 3,3a | 1 Day Postoperative | 1-2 days postoperative* | 3,3a |
| 4 | 1 Month Postoperative | 30 (±10) days postoperative** | 4 |
| 5 | 3 Months Postoperative | 90 (±20) days postoperative** | 5 |

<sup>\*</sup> relative to the operative eye

# 9.2.1. Preoperative

At the preoperative exam, subjects will be consented, qualified for the study (compared with inclusion/exclusion criteria), and assigned a study ID/subject number. Subject numbers will be assigned sequentially at each site in the order of enrollment. Pre-operative qualification should take place no more than 30 days prior to surgery.

A medical history will be taken and exams will include the tests described below:

- manifest refraction,
- visual acuity
- preoperative QUVID questionnaire
- preoperative IOLSAT questionnaire

In addition, all site-specific, routine, usual standard of care preoperative measures should be undertaken.

Measurements should be made as described in section 9.3 below.

#### 9.2.2. Operative (Surgery)

All subjects will undergo cataract surgery with implantation of the Clareon PanOptix IOL. The surgeon's usual standard of care with regard to treatment and medication will be used for all study subjects. Surgery planning and IOL power calculation will be performed using the surgeon's preferred method, with an initial a-constant provided by Alcon. If a toric IOL is used, planning will be performed with the Alcon Toric calculator that takes the effects of posterior corneal astigmatism into account.

<sup>\*\*</sup> relative to the date the last eye is operated on

Surgical findings will be recorded and any adverse events/serious adverse events

(AEs/SAEs) occurring during surgery will be noted at this visit. Any other problems during surgery and comments regarding surgery will be documented.

Any subject whose surgery is not completed successfully will be documented in the appropriate case report form. These subjects will be monitored for safety but clinical performance data may be excluded from the analysis.

# 9.2.3. Postoperative 1 Day

All routine, usual standard of care postoperative measures should be undertaken. In addition, the subject will undergo VA and lens orientation testing in accordance with the specifications below (Section 9.3). Adverse events will be monitored.

# 9.2.4. Postoperative 1 Month

All routine, usual standard of care postoperative measures should be undertaken. In addition, the subject will undergo a manifest refraction, VA, and lens orientation testing and complete the QUVID and IOLSAT questionnaires (Section 9.3). Any device deficiencies or adverse events will be monitored.

# 9.2.5. Postoperative 3 Months

All routine, usual standard of care postoperative measures should be undertaken. In addition, the subject will undergo a manifest refraction, VA, and lens orientation testing and complete the QUVID and IOLSAT questionnaires (Section 9.3). Any device deficiencies or adverse events will be monitored.

### 9.2.6. Exit Procedures

In the event of premature exit from the study, all study related examinations should be completed where possible. The Exit CRF should be completed, noting that the subject did not complete the study and the reason for premature study exit. If no premature exit from the study occurs, the Exit CRF should be completed at the end of Visit 5 (Postoperative 3 Months).

#### 9.3. Study Methods and Measurements

All routine testing and basic eye examinations should be carried out at each study visit. Abnormalities should be recorded in the CRF "Comment" section. Specific study examination procedures are outlined below.

#### 9.3.1. Manifest Refraction

Perform a manifest refraction with a high contrast logMAR chart under photopic lighting conditions (>85 cd/m<sup>2</sup>). Document refraction results with sphere, cylinder and axis readings. If uncorrected visual acuity is not improved by

manifest refraction, use zero for sphere and cylinder and draw a line through the blank for the axis.

*Note:* Each subject should be manually refracted to his/her best correction by an ophthalmologist, optometrist, or a skilled technician using a phoropter or trial lenses.

# 9.3.2. Visual Acuity (VA)

Visual acuity will be measured using the M&S Technologies Clinical Trial System. All relevant data will be recorded internally.

It is sufficient to record the uncorrected VA at distance only for the 1-day visit.

All other visual acuity testing is performed binocularly. Postoperatively conduct testing uncorrected at all visits. In addition, conduct testing with the manifest distance refraction in place at 1 month and 3 months post-operatively.

#### Distance VA

Measure distance VA at a distance of 6 m.

#### Intermediate VA

Measure intermediate VA at a distance of 60 cm.

#### Near VA

Measure near VA at a distance of 40 cm or 33 cm.

#### 9.3.3 Questionnaires

The patient satisfaction (IOLSAT) questionnaire and the visual disturbance (QUVID) questionnaire, related to quality of vision, will be administered to subjects at the 1 and 3-month visits. The administrator should ensure the subjects understand the nature of the questions but should not interpret them for the subject.

#### 9.4. Unscheduled Visits

Unscheduled exams may be conducted at the discretion of the Investigator with all relevant information from the exam recorded in the source documents and on the Unscheduled Visit pages within the CRF booklet.

### 9.5. Discontinued Subjects

Discontinued subjects are those who do not have an exit visit or who come into the office to be exited prior to the scheduled final study visit. Subjects may be discontinued from the study at any time if, in the opinion of the investigator, their continued participation in the study poses a risk to their health. The reasons for discontinuation include:

a. Adverse event;

- b. Lost to follow-up;
- c. Subject decision unrelated to an adverse event;
- d. Protocol violation;
- e. Treatment failure;
- f. Other.

To ensure the safety of all subjects who discontinue prior to Visit 5, investigators should assess each subject and, if necessary, advise them of any therapies and/or medical procedures that might be needed to maintain their health. Any changes in medical health and/or use of concomitant medications should also be captured.

#### 10. ANALYSIS PLAN

#### 10.1. Analysis Data Sets

All subjects who are enrolled in the study will be evaluated for safety. Efficacy analyses will be performed based on data from those eyes where uncomplicated cataract surgery with PanOptix IOL implantation was completed.

#### 10.2. Statistical Methodology

A summary of the data will be prepared for all measurement time points. Summaries of the changes observed between the 1-month and 3-month post-operative visits will also be summarized.

For variables measured on a continuous scale, these summaries will include the sample size, as well as the mean, standard deviation, median, minimum, and maximum. For variables measured on a categorical scale, summaries will provide the number and percentage of subjects who provided each score (or change in scores). These summaries will be provided for all eyes completing the study.

#### 10.2.1. Within-treatment Changes

For variables measured on a continuous scale, the statistical significance of within-treatment changes between time points will be investigated using paired t-tests. For variables measured on an ordinal categorical scale, the Wilcoxon signed-rank test will be employed.

#### 10.3. General Statistical Considerations

The statistical analyses will be performed using R, version 4.1.2 or higher. Any statistical tests of hypotheses will employ a level of significance of alpha=0.05.

# 11. SAMPLE SIZE JUSTIFICATION

There is no particularly relevant sample size justification with a single-arm study. It is worth noting that prior studies with between 30 and 35 subjects in any given study group have allowed successful distinctions to be made in the performance of different trifocal IOLs, including PanOptix.<sup>3</sup> It is expected that 32 subjects (64 eyes) will provide sufficient data to characterize the clinical performance of the lens. To allow for 10% dropout, 35 subjects (70 eyes) will be enrolled.

#### 12. CONFIDENTIALITY/PUBLICATION OF THE STUDY

The existence of this Study is confidential and should not be discussed with persons outside of the Study. Results will be submitted for publication and presentation at national and/or international meetings. A manuscript will be submitted to peer-review journals for publication but there is no guarantee of acceptance.

All study data will be collected on appropriate Case Report Forms (CRFs). No protected health information will be included on the forms. CRFs will be retained in the patient's file for a minimum period of 3 years. Collected information will only be used for purposes of this study and no information will be sold to third parties. The following people will have access to your study records:

- Study Doctor and staff involved with the study
- Study Monitor or Auditor
- Sponsor Company or Research Institution
- Review boards or accrediting agencies
- Other State or Federal Regulatory Agencies

The de-identified data may be shared with other researchers for future analysis.

#### 13. QUALITY COMPLAINTS AND ADVERSE EVENTS

All subjects will be monitored for adverse events over the course of the study. A place to record any adverse event is included on each case report form.

# 13.1. General Information

An Adverse Event (AE) is any untoward medical occurrence in a subject who is administered. a study treatment regardless of whether or not the event has a causal relationship with the treatment. An AE, therefore, can be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment. In clinical studies, an AE can include an untoward medical occurrence occurring at any time, including run-in or washout periods, even if no study treatment has been administered.

#### 13.2. Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the Investigator should inquire about AEs by asking if the patient has any problems.

#### 13.3. Procedures for Recording and Reporting AEs and SAEs

Subsequent to signing an informed consent form, all untoward medical occurrences that occur during the course of the study must be documented on an Adverse Event Form

7 July 2022

(AEF). A separate AEF must be filled out for each event. When possible, signs and symptoms indicating a common underlying pathology should be documented as one comprehensive event. For each recorded event, the AE documentation must include the onset date, outcome, resolution date (if event is resolved), intensity (i.e., severity), any action with study treatment taken as a result of the event, and an assessment of the adverse event's relationship to the study treatment.

#### **Nonserious Adverse Events**

A nonserious AE is defined as any untoward change in a subject's medical health that does not meet serious criteria noted below (e.g., is not life-threatening, does not require hospitalization, does not prolong a current hospitalization, is not disabling, etc.). All adverse events must be reported regardless of whether or not they are related to the study treatment.

For nonserious adverse events, an AEF containing all available information will be collected on a routine basis and submitted to the Medical Monitor at the close of the study.

#### **Serious Adverse Events**

A serious adverse event (SAE) is defined as any adverse experience that meets any of the following criteria:

- Results in death.
- Is life-threatening.

NOTE: Life-threatening means that the subject was at immediate risk of death from the reaction as it occurred; i.e., it does not include a reaction which hypothetically might have caused death had it occurred in a more severe form.

- Requires inpatient hospitalization or prolongation of existing hospitalization. NOTE: In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious.
- Results in persistent or significant disability/incapacity. Disability is defined as a substantial disruption of a person's ability to conduct normal life functions.

  NOTE: The term disability means a substantial disruption of a person's ability to conduct normal life functions. This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, or accidental trauma (e.g., sprained ankle) which may interfere or prevent everyday life functions but do not constitute a substantial disruption.
- Is an important medical event. An important medical event is an event that may not result in death, be life-threatening, or require hospitalization but may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the subject and may require medical or surgical intervention to prevent one of the

outcomes listed in the definitions for SAEs. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in subject hospitalization, or the development of drug dependency or drug abuse.

All available information on a serious adverse event(s) and any other associated AE, if applicable, must be forwarded to the study coordinator for forwarding to the Medical Monitor immediately (i.e., within one working day of the Investigator's or site's knowledge of the event) as follows:

- In studies utilizing EDC (electronic data capture), all available information for the SAE and any associated AE(s) must be entered immediately into the EDC system.
- Additional information for any applicable event is to be reported as soon as it becomes available.

In addition to the reporting of serious adverse events to the study Medical Monitor, the SAE must be reported to the IRB / IEC according to their requirements.

The investigator must document all adverse device events (serious and nonserious but related) and all serious adverse events (related and unrelated) on the Adverse Device Effect and Serious Adverse Event Form. Any device quality complaints will also be documented.

- Both the Quality Complaint Form and the Adverse Device Effect and Serious Adverse Event Form must be e-mailed immediately to the study coordinator.
- Additional relevant information is to be reported as soon as it becomes available.

Study coordinator contact information is provided below.

Table 13.3.-1: Contact Information for the Study

| Study Staff<br>(Coordinator) | <b>Business Phone</b> | e-mail | 24-hour<br>Office Phone |
|---|---|---|---|
| Jamie Dixon | 863-385-1544 | j.dixon@newsomeye.net | 863-385-1544 |

Further, depending upon the nature of the adverse event (serious or nonserious) or quality complaint being reported, the study sponsor may request copies of applicable portions of the subject's medical records. The investigator must also report all adverse events and quality complaints according to the relevant IRB requirements.

# 12.3.1 Intensity and Causality Assessments

For every adverse event and quality complaint, the investigator must assess the causality as Related or Not Related to the medical device under investigation. An assessment of causality will also be performed by the Medical Monitor utilizing the same definitions, as shown below:

# **Causality**

Related An adverse event or quality complaint classified as related may be

either definitely related or possibly related where a direct cause and effect relationship with the medical device has not been demonstrated, but there is a reasonable possibility that the adverse event or quality complaint was caused by the medical device.

Not Related An adverse event or quality complaint classified as not related may

either be definitely unrelated or simply unlikely to be related (i.e., there are other more likely causes for the adverse event or quality

complaint).

Where appropriate, the investigator must assess the intensity (severity) of the adverse event as mild, moderate, or severe based on medical judgment with consideration of any subjective symptom(s), as defined below:

# Intensity (Severity)

Mild An adverse event is mild if the subject is aware of but can easily

tolerate the sign or symptom.

Moderate An adverse event is moderate if the sign or symptom results in

discomfort significant enough to cause interference with the

subject's usual activities.

Severe An adverse event is severe if the sign or symptom is incapacitating

and results in the subject's inability to work or engage in their

usual activities.

The investigator must document any action taken (i.e., medication, intervention, or treatment plan) and outcome of the adverse event or quality complaint when applicable.

#### 13.4. Follow-Up of Adverse Events and Quality Complaints

The investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study. Any additional data from these follow-up procedures must be documented and available to the study coordinator who, with the Medical Monitor, will determine when the data need to be documented on the CRFs.

# 13.5. Safety Analyses

The type, severity, duration and frequency of reported ocular adverse events will be tabulated. Adverse events will also be summarized for events that were considered treatment-related.

#### 14. GCP, ICH and ETHICAL CONSIDERATIONS

This study will be conducted in compliance with Good Clinical Practices (GCPs), including International Harmonization (ICH) Guidelines, and in general, consistent with the 1996 version of the Declaration of Helsinki. In addition, all applicable local, state and federal requirements will be adhered to.

This study is to be conducted in accordance with Institutional Review Board regulations. The investigator will obtain appropriate IRB/ethics committee approval prior to initiating the study.

The study will be registered with clinicaltrials.gov.

# 14.1 Confidentiality

The data collected will be data typical for the procedure(s) when performed on eyes outside the study. Any data collected will become part of the patient's clinical record. The data will be subject to the same privacy and confidentiality as other data in the clinical record.

Only the principal investigator, research consultant and clinic staff will have access to the data collected. All data shared outside the practice will be de-identified; patients' protected health information will not be available and will not be reported in any analyses or publications. No data will be sold to third parties. De-identified data may be used for future research.

#### 15. STANDARD EVALUATION PROCEDURES

Table 15.1. Proposed Visits and Study Assessments

(visits are by patient, with both eyes tested)

| Activity | Pre-<br>operative | Operative | | Postoperativ | e |
|---|---|---|---|---|---|
| | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 |
| | | | 1 Day | 1 Month | 3 Months |
| Informed Consent | Χ | | | | |
| Demographics | Х | | | | |
| General Information:<br>Medical History | Х | | | | |
| Surgery | | X | | | |
| Manifest refraction | Х | | | Х | Х |
| Monocular uncorrected distance VA (6m) | Х | | Χ | Х | Х |
| Monocular corrected distance VA (6m) | Х | | | Х | Х |
| Binocular uncorrected and best-<br>corrected distance VA (6m) | | | | Х | Х |
| Binocular uncorrected and best distance-corrected intermediate VA (60cm) | | | | Х | X |
| Binocular uncorrected and best distance-corrected near VA (40cm & 33cm) | | | | Х | Х |
| Binocular Distance Corrected Defocus Curve (6m) | | | | | Х |
| IOLSAT Patient Satisfaction Survey | Х | | | | Х |
| QUVID Visual Disturbance questionnaire | Х | | | | Х |
| Monitor for Adverse Events and Device Deficiencies | | Х | Х | Х | Х |
| Complete Exit Form <sup>1</sup> | | | | | Х |

<sup>&</sup>lt;sup>1</sup> Complete Exit Form upon termination of subject participation, or at Visit 5, whichever occurs first.

#### 16. DATA CONFIDENTIALITY

No protected health information (PHI), including the patient's name and date of birth, will be collected; to ensure this, no PHI information is permitted to be entered on any of the Case Report Forms (CRFs). Subjects will only be identified by subject IDs and identities will be removed at the initial visit so that there is no further need to protect or destroy the information. Collected information will only be used for purposes of this study and no information will be sold to third parties. The non-PHI information collected may be used for future research, though there is currently no plan to do so.

# 17. FINANCIAL AND INSURANCE INFORMATION/STUDY RELATED INJURIES

Every effort to prevent study-related injury will be taken by the Study Doctor and staff. In the event a patient is injured as a direct result of the study while following the Study Doctor's instructions and the study requirements, the patient will be instructed to contact his or her doctor immediately. The Study Doctor is to treat the injured subject as needed for those injuries caused directly by this research study. In the event of injury or illness caused by or occurring during a subject's participation in this research study, all charges for medical care provided to the subject will be billed to his or her insurance company. The Study Doctor or Sponsor does not offer to cover the medical care costs for injuries or illnesses that are not caused directly by the research study. The Sponsor does not offer to provide any other compensation, unless specifically agreed to elsewhere in this document. This information will be provided to each study subject before the start of the study in the consent form.

#### 18. STUDY ENDPOINT CRITERIA

# 18.1. Patient Completion of Study

If a study patient has completed the final visit (Visit 5) of the study, he/she is considered to have completed the study.

#### 18.2. Patient Discontinuation

Each study patient may voluntarily discontinue the study at any time they choose. Study patients who cannot complete the study for administrative reasons (e.g., non-compliance, failure to meet visit schedule, etc.) will be discontinued from the study. Study patients discontinued during the enrollment phase (prior to surgery) of the study will be replaced.

#### 18.3. Patient Termination

A study patient will be terminated if the study patient develops any severe adverse event that may be related to the study. A study patient will receive appropriate treatment at the discretion of the investigator. Notification of termination will be clearly documented. These study patients are considered to have completed the study and will not be replaced.

#### 18.4. Study Termination

The investigator with appropriate notification may terminate the study. If, after clinical observations, the investigator feels that it may be unwise to continue the study, he may stop the study.

#### 18.5. Study Completion

The study will be complete when all enrolled patients have completed Visit 5 or have been terminated from the study.

#### 19. SUMMARY OF RISKS AND BENEFITS

# 19.1. Summary of risks

The risks with this study are similar to those for any patient electing multifocal IOLs.<sup>1-3</sup> There is no increased risk associated with the proposed study.

# 19.2. Summary of benefits

Studies of trifocal IOLs have demonstrated that patients are likely to have relatively good distance, intermediate, and near vision.<sup>1-3</sup>

Subjects may be compensated up to \$600 for completing the study.

#### **REFERENCES**

- 1. Blaylock JF, Hall B. Clinical outcomes of a diffractive trifocal intraocular lens with femtosecond laser, digital tracking, and intraoperative aberrometry. *Can J Ophthalmol.* 2021.
- 2. Blaylock JF, Hall B. Astigmatic results of a diffractive trifocal Toric IOL following intraoperative aberrometry guidance. *Clin Ophthalmol.* 2020;14:4373-4378.
- 3. Alio JL, Plaza-Puche AB, Alio Del Barrio JL, et al. Clinical outcomes with a diffractive trifocal intraocular lens. *Eur J Ophthalmol.* 2018;28(4):419-424.